CLINICAL TRIAL: NCT06172023
Title: Evaluation of Antimicrobial Efficacy and Postoperative Pain After Using Silver Nanoparticles and Chitosan Nanoparticles Against Enterococcus Faecalis and Candida Albicans Biofilm (An in Vitro - in Vivo Study)
Brief Title: Evaluation of Antimicrobial Efficacy and Postoperative Pain After Using Silver Nanoparticles and Chitosan Nanoparticles Against Enterococcus Faecalis and Candida Albicans Biofilm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahmed Amr El Wakad, Doctorate candidate at the Faculty of Dentistry, Minia University, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: (RHDIRB2017122004) (438)
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Endodontic Disease
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Silver Nanoparticles Irrigant (Experimental)
  Interventions: Drug: Silver Nanoparticles Irrigant
- Chitosan Nanoparticle Irrigant (Experimental)
  Interventions: Drug: Chitosan Nanoparticles Irrigant
- 2.6% NaOCl and 17% EDTA sol (Active Comparator)
  Interventions: Drug: Silver Nanoparticles Irrigant; Drug: Chitosan Nanoparticles Irrigant

INTERVENTIONS:
Drug: Silver Nanoparticles Irrigant — Nanosilver irrigant solution
  Arms: 2.6% NaOCl and 17% EDTA sol; Silver Nanoparticles Irrigant
Drug: Chitosan Nanoparticles Irrigant — Chitosan nanoparticles irrigant solution
  Arms: 2.6% NaOCl and 17% EDTA sol; Chitosan Nanoparticle Irrigant

SUMMARY:
Silver nanoparticles possess unique physicochemical and biological properties in addition to their antibacterial capabilities. Similarly, zinc oxide nanoparticles have demonstrated antibacterial effects against a wide range of bacteria, including heat and pressure resistant spores. Given these characteristics, it would be valuable to evaluate and compare a new irrigation solution containing nanosilver and nanozinc-oxide particles with sodium hypochlorite. Furthermore, Chitosan Nanoparticles are expected to exhibit enhanced antibacterial activity compared to regular-sized Chitosan due to their ability to penetrate and disrupt microbial cell membranes. Consequently, the current study aims to assess and compare the antibacterial activity of Silver Nanoparticles and Chitosan Nanoparticles, as well as their impact on post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable healthy patients (category: American society of anesthesiologists class I).
* The patient ranges in age from 20 to 40.
* No sexual orientation
* Necrotic pulp evaluated by thermal or electrical pulp testing.
* Enough crown structure to provide adequate isolation.
* One root and one canal.
* Patients' desire to engage in this research.
* Patients' comprehension of the visual analogue scale (VAS).
* Patients' ability to sign informed consent.

Exclusion Criteria:

* Endodontic treatment for the tooth previously.
* Teeth with poor conditions for using rubber dams.
* Vital pulp tissue was observed throughout the treatment.
* Patients who have a medical condition.
* Teeth with open apices that are immature
* Women who are pregnant or breastfeeding.
* Psychologically disturbed patients.
* Patients having a history of allergy to any of the research drugs were barred from participation.
* A periodontally affected tooth with grade 2 or 3 mobility.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Assessment | 6, 12, 24, 48, and 72 hours
  Each patient was given a pain scale chart (VAS scale) before every endodontic operation to record his or her pain level. The VAS is a 10-point scale with values ranging from 0 to 10, with 0 representing "No pain," (1-3) representing "mild pain," (4-6) representing "moderate pain," and (7-10) representing "worst imaginable pain." At 6, 12, 24, 48, and 72 hours, each patient was instructed to use the VAS scale (0-10) to rate the presence and severity of discomfort after obturation.

SECONDARY OUTCOMES:
Antimicrobial Activity Assessment | 1 hour, 24 hours, 7 days, and 30 days
  A sterile paper point was placed in each root canal to a level roughly 1 mm short of the apex, depending on working length radiographs, to get a sample from the root canal. The samples were suspended in a suspension of 25 microliters, which was pipetted onto a BHI agar plate. The colonies were counted using a Reichert-Jung colony counter after 1 hour, 24 hours, 7 days, and 30 days of incubation at 37oC in an anaerobic jar.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided